CLINICAL TRIAL: NCT03880955
Title: A Post-Market Clinical Evaluation of the ReUnion Reverse Shoulder Arthroplasty (RSA) System
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision to stop at 2 year follow-up
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: ReUnion RSA Study
Record Dates: First submitted 2019-03-07; First posted 2019-03-19 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ReUnion RSA System: Subject's joint has gross rotator cuff deficiency, a functional deltoid muscle and is anatomically and structurally suited to receive the implant and subject has one or more of the following:
  * Painful, disabling joint disease of the shoulder resulting from degenerative arthritis or rheumatoid arthritis
  * Failed previous shoulder joint replacement
  Interventions: Device: ReUnion RSA System

INTERVENTIONS:
Device: ReUnion RSA System — The ReUnion RSA System is designed as a reverse total shoulder endoprosthesis to address unrepairable gross rotator cuff tear, rotator cuff arthropathy with pseudoparalysis of the shoulder joint, advanced arthritic and rheumatic disorders affecting the shoulder joint, and failed previous shoulder arthroplasty. The ReUnion RSA System is comprised of a Humeral Cup, Humeral Insert, Glenosphere, Glenoid Baseplate and Screws. The intended purposes of the ReUnion RSA System are to achieve pain relief, improvement of range of motion and restoration or improvement of the shoulder function while ensuring long-term replacement of the shoulder joint with sufficient stability of all endoprosthesis components.

SUMMARY:
This investigation is a prospective, multicenter clinical investigation. It is anticipated that a total of eighty (80) subjects will be enrolled at approximately 4-7 sites. The clinical investigation has been designed to follow the surgeon's standard of care for joint arthroplasty subjects, which entails clinical evaluation on a regular ongoing basis, or as needed should the subject become symptomatic in the treated joint.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to demonstrate the safety and efficacy/performance of the ReUnion RSA System. Efficacy/performance of the procedure will be measured the American Shoulder and Elbow Surgeons (ASES) Shoulder Score. Safety of the ReUnion RSA System will be demonstrated through reporting of device-related intra-operative and post-operative Adverse Events (AEs). Enrolled subjects will be assessed at Pre-Operative, Operative/Discharge, and at 6 Weeks, 6 Months, 12 Months, 24 Months and annually thereafter up to 10 years following the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign the informed consent.
* Subject is willing and able to comply with postoperative scheduled clinical and radiographic evaluations.
* Subject is male or non-pregnant female and 18 years or older at the time of surgery.
* Subject's joint has gross rotator cuff deficiency, a functional deltoid muscle and is anatomically and structurally suited to receive the implant and subject has one or more of the following:

  * Painful, disabling joint disease of the shoulder resulting from degenerative arthritis or rheumatoid arthritis
  * Failed previous shoulder joint replacement

Exclusion Criteria:

* Subject has an active or suspected latent infection in or about the shoulder joint.
* Subject has mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure or complications in postoperative care.
* Subject has bone stock compromised by disease, infection or prior implantation which cannot provide adequate support and/or fixation to the prosthesis.
* Subject has anticipated activities which would impose high stresses on the prosthesis and its fixation.
* Subject is obese such that he/she produces a load on the prosthesis which can lead to failure of fixation of the device or to failure of the device itself.
* Subject has concomitant disease(s) which may significantly affect the clinical outcome.
* Subject has traumatic or pathologic fracture of the proximal humerus

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 80 subjects are to be enrolled in this clinical investigation. The clinical investigation has been designed to follow the surgeon's standard of care for joint arthroplasty subjects, which entails clinical evaluation on a regular ongoing basis, or as needed should the subject become symptomatic in the treated joint.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma and Extremities
Locations (3):
- United States (3):
  - Great Plains Orthopedics, Peoria, Illinois
  - Steadman Hawkins Clinic of the Carolinas, Greenville, South Carolina
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ReUnion RSA System: Subject's joint has gross rotator cuff deficiency, a functional deltoid muscle and is anatomically and structurally suited to receive the implant and subject has one or more of the following:
  * Painful, disabling joint disease of the shoulder resulting from degenerative arthritis or rheumatoid arthritis
  * Failed previous shoulder joint replacement
  ReUnion RSA System: The ReUnion RSA System is designed as a reverse total shoulder endoprosthesis to address unrepairable gross rotator cuff tear, rotator cuff arthropathy with pseudoparalysis of the shoulder joint, advanced arthritic and rheumatic disorders affecting the shoulder joint, and failed previous shoulder arthroplasty. The ReUnion RSA System is comprised of a Humeral Cup, Humeral Insert, Glenosphere, Glenoid Baseplate and Screws. The intended purposes of the ReUnion RSA System are to achieve pain relief, improvement of range of motion and restoration or improvement of the shoulder function while ensuring long-term replacement of the shoulder joint with sufficient stability of all endoprosthesis components.
Period: Overall Study
Arm/Group | ReUnion RSA System
Started | 102
Completed | 57
Not Completed | 45
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 12
Not completed — Withdrawal by Subject | 4
Not completed — Missing- Study Site Closed | 27

BASELINE CHARACTERISTICS:
Arm/Group | ReUnion RSA System
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.80 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Black or African | 6
  Ethnicity: Caucasian | 92
  Ethnicity: Other | 4
Region of Enrollment [Number; unit: participants]
  United States | 102
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 29.49 (5.13)

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder and Elbow Surgeons (ASES) Shoulder Score
Description: This is a mixed outcome reporting measure, applicable for use in patients with shoulder pathology regardless of diagnosis and consists of a pain visual analog scale (VAS) and 10 functional questions. The primary endpoint of the clinical investigation is to demonstrate non-inferiority of the device to the selected literature controls, as measured by the ASES Shoulder Score at 24 Months post-operative. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Time Frame: 24 Months
Population: 54 out of 102 Subjects had available data at 24mths.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ReUnion RSA System
Number analyzed (Participants) | 54
units on a scale | 88.19 (15.39)

2. Secondary Outcome: Safety Will be Measured by Capturing the Incidence Rate of Device-related Intra-operative Adverse Events.
Description: Secondary outcome measures to assess safety by capturing the incidence rate of device-related intra-operative adverse events.
Time Frame: 24 months
Population: 4 out of 102 Subjects with reportable Intra-operative Adverse Events. Please see Adverse Events section for break-down.
Measure: Count of Participants; unit: Participants
Arm/Group | ReUnion RSA System
Number analyzed (Participants) | 102
Participants | 4

3. Secondary Outcome: Safety Will be Measured by Capturing the Incidence Rate of Device-related Post-operative Adverse Events.
Description: Secondary outcome measures to assess safety by capturing the incidence rate of device-related post-operative adverse events.
Time Frame: 24 months
Population: 16 out of 102 Subjects with reportable post-operative Adverse Events. Please see Adverse Events section for break-down.
Measure: Count of Participants; unit: Participants
Arm/Group | ReUnion RSA System
Number analyzed (Participants) | 102
Participants | 16

4. Secondary Outcome: Efficacy Will be Measured by Monitoring All Implant Survivorship in All Subjects Who Have the Reverse Total Shoulder Endoprosthesis With the ReUnion RSA System.
Description: Secondary outcome measures to assess efficacy by monitoring all implant survivorship in all subjects who have the reverse total shoulder endoprosthesis with the ReUnion RSA System.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | ReUnion RSA System
Number analyzed (Participants) | 102
Participants | 101

ADVERSE EVENTS:
Time Frame: 24 months
Description: Procedural and device related events will be described and collected on the AE form. It is the responsibility of the operating surgeon/s to be aware and note the adverse effects from the package insert/instructions for use by the manufacturer/sponsor.
Arm/Group | ReUnion RSA System
All-Cause Mortality (participants affected / at risk) | 1/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 20/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReUnion RSA System (N=102)
Deep infection (Infections and infestations) | 2
Heterotopic ossification, asymptomatic (Musculoskeletal and connective tissue disorders) | 5
Heterotopic ossification, symptomatic (Musculoskeletal and connective tissue disorders) | 2
Intraoperative fracture of the glenoid (Musculoskeletal and connective tissue disorders) | 1
Intraoperative fracture of the humerus (Musculoskeletal and connective tissue disorders) | 1
Late infection (e.g. hematogenous or protracted) (Infections and infestations) | 1
Pain related to the implant, severe (Product Issues) | 1
Radiographic lucency, humeral (Musculoskeletal and connective tissue disorders) | 2
Stress fracture of the acromion or the scapular neck (Musculoskeletal and connective tissue disorders) | 3
Wound complications (e.g. hematoma, wound healing disturbances) (Skin and subcutaneous tissue disorders) | 1
Other (inferior osteophyte off of glenoid) (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The protocol allowed for subjects to be assessed annually up to 10 years after the index procedure, but the study was closed early and collected assessments only through 24 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT03880955/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT03880955/SAP_001.pdf